CLINICAL TRIAL: NCT05750186
Title: The Effect of Abdominal Massage Applied After Surgery on Gastrointestinal Symptoms and Comfort Level
Brief Title: The Effect of Abdominal Massage Applied After Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Semiha Kurt, Research Assistant, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Skurt-AbMa-01
Record Dates: First submitted 2023-02-03; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Reflux, Gastroesophageal; Abdominal Pain; Constipation; Diarrhea; Dyspepsia
Keywords: Abdominal Massage; Postoperative Care; Nonpharmacological Methods; Independent Nursing Practices
MeSH Terms: conditions — Gastroesophageal Reflux; Abdominal Pain; Constipation; Diarrhea; Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal Massage Group (Experimental): At the first encounter with the patient; Patient Information Form, Gastrointestinal Symptom Rating Scale, General Comfort Scale and Functional Independence Scale will be applied.
  * From the morning of the first day, abdominal massage will be applied to the patients 2 times a day, in the morning and in the evening, for 3 days (15 minutes).
  * Then, applying abdominal massage to the patients in the experimental group. After each massage application, the patient's bowel sounds/movements will be listened to.
  * Medicines such as laxatives, suppositories and enemas will not be given to the experimental group and Bristol Stool Scale will be filled in for patients who defecate within this period.
  * In order to evaluate the abdominal massage and its effect on the comfort level of the patients, the Gastrointestinal Symptom Rating Scale, General Comfort Scale and Functional Independence Scale will be applied again at the end of the 3rd day after the application of abdominal massage.
  Interventions: Other: Abdominal Massage
- Control Group (No Intervention): * Patients who did not defecate within the first 3 days after surgery will constitute the control group.
  * At the first encounter with the patient; A Patient Information Form, Gastrointestinal Symptom Rating Scale (GSS), General Comfort Scale (GAS) and Functional Independence Scale (FIM) will be administered.
  * From the first encounter, patients will be given medications that are in line with their clinical routine, such as laxatives, suppositories and enemas, according to the doctor's request.
  * Intestinal sounds/movements of the patients will be listened to 6 times, 2 times a day for 3 days.
  * Bristol Stool Scale will be filled in for patients who defecate within this period.
  * At the end of the 3-day follow-up of the patients, Gastrointestinal Symptom Rating Scale, General Comfort Scale and Functional Independence Scale will be applied again and the first stool of the patients who defecate will be evaluated with the Bristol Stool Scale.

INTERVENTIONS:
Other: Abdominal Massage — Abdominal massage is a noninvasive application that stimulates bowel movements by applying patting, kneading and vibration movements over the abdominal wall to the area where the intestines are located. It increases peristalsis, creates a mechanical and reflex effect on the intestines, reducing the individual's feeling of pain and discomfort.
  Arms: Abdominal Massage Group

SUMMARY:
This research is carried out by research assistant Semiha Kurt under the supervision of Associate Professor Nuray TURAN.

In this research aimed to examine the effect of abdominal massage applied after surgical ıntervention on gastrointestinal symptoms and comfort level. The type of this study designed as randomized controlled experimental. The research hypotheses are as follows; H1: Abdominal massage applied after surgery reduces the gastrointestinal symptoms of patients.

H2: Abdominal massage applied after surgery increases the comfort level of patients.

The population of the research will consist patients who were hospitalized and underwent surgical intervention between January 2023 and July 2024 in the Orthopedics and Traumatology Clinic of the Istanbul Medical Faculty Hospital in Istanbul.The sample of the research will consist patients who cannot defecate for 3 days after surgery and who meet other sample selection criteria.

As a result of the power analysis (G*Power 3.0.10); at least 34 samples found to be sufficient for each group with f=0.20 effect size, 90% power and 5% margin of error (n1:34, n2:34). The number of samples determined as 68 (including the experimental and control groups).

Data will be collected through the Patient Information Form, Bristol Stool Scale, Gastrointestinal Symptom Rating Scale, General Comfort Scale, and Functional Independence Scale. The patient information form was prepared by the researchers in line with the literature. Permission was obtained from the scale owners for the scales to be used in the study.

In the implementation phase of the research; in the formation of the experimental and control groups, the assignment of the patients to the experimental and control groups will be provided by randomization in the computer. Abdominal massage will be applied to the patients in the experimental group twice a day, in the morning and evening, for 3 days. Each abdominal massage will be applied for 15 minutes. The routine practice of the clinic will continue in the patients in the control group.

Institutional permission from Istanbul Medical Faculty and ethics committee approval (Number: E-74555795-050.01.04-412448) from Istanbul University-Cerrahpasa Non-Interventional Research Ethics Committee obtained in order to conduct the study. Statistical analysis of research data will be done using a package program called SPSS (IBM SPSS Statistics 24). The expenses of the research will be covered by the researcher.

DETAILED DESCRIPTION:
Gastrointestinal symptoms that cause discomfort in patients and reduce their quality of life and comfort include disorders related to the esophagus, stomach, duodenum, jejunum, ileum, large intestine, sigmoid colon and rectum. These symptoms: reflux, abdominal pain, constipation, diarrhea and indigestion. After surgery, slowing of gastrointestinal system motility and change in eating habits can cause serious problems in patients by causing the development of gastrointestinal symptoms such as post-operative nausea, vomiting and hiccups. The development of these symptoms, on the other hand, prolongs the hospital discharge time of patients and may lead to increased costs. Prolonged persistence of abdominal distension after surgery; It may cause delayed wound healing due to increased pressure in the incision area, deep vein thrombosis in the legs due to decreased venous return, paralytic ileus and gastric dilation due to decreased blood flow in the intestine.Constipation; It can cause pain, nausea, vomiting, distention, feeding intolerance and contribute to the development of intestinal obstruction or perforation if not treated. There are many care and treatment methods, including pharmacological and non-pharmacological, stimulating gastrointestinal motility after surgical intervention. Abdominal massage, which is one of the non-pharmacological methods, is an important intervention in the management of gastrointestinal symptoms. Abdominal massage is a noninvasive application that stimulates bowel movements by applying patting, kneading and vibration movements over the abdominal wall to the area where the intestines are located. It increases peristalsis, creates a mechanical and reflex effect on the intestines, reducing the individual's feeling of pain and discomfort. The aim in the management of gastrointestinal symptoms is to prevent problems that may develop and to increase the quality of life and comfort of the patient by reducing these problems when they occur. Nurses are one of the team members who can diagnose and communicate with all aspects of healthy/sick individuals and their families, and take an active role in the management of gastrointestinal symptoms that may develop after surgical intervention and in the care of the individual. In this context, nurses have important roles and responsibilities. When the literature is examined, it has been observed that patients experience various problems related to gastrointestinal symptoms after surgical intervention. Abdominal massage, which is one of the non-pharmacological methods, is one of the most important independent nursing interventions in the management of gastrointestinal symptoms, as it is low cost and effective, without side effects for healthy/sick individuals and their families. In this context, this study planned to determine the effect of abdominal massage applied to patients after surgical intervention on gastrointestinal symptoms and comfort level.

In this research aimed to examine the effect of abdominal massage applied after surgical ıntervention on gastrointestinal symptoms and comfort level. The type of this study designed as randomized controlled experimental. The research hypotheses are as follows; H1: Abdominal massage applied after surgery reduces the gastrointestinal symptoms of patients.

H2: Abdominal massage applied after surgery increases the comfort level of patients.

The independent variables of the study the application of abdominal massage, the individual and disease characteristics of the patients; dependent variables are gastrointestinal symptom and comfort level scores.

The research will be carried out in the Orthopedics and Traumatology Clinic of Istanbul Medical Faculty Hospital in Istanbul between January 2023 and July 2024.

The population of the research will consist patients who were hospitalized and underwent surgical intervention between January 2023 and July 2024 in the Orthopedics and Traumatology Clinic of the Istanbul Medical Faculty Hospital in Istanbul.The sample of the research will consist patients who cannot defecate for 3 days after surgery and who meet other sample selection criteria.

Data will be collected through the Patient Information Form, Bristol Stool Scale, Gastrointestinal Symptom Rating Scale, General Comfort Scale, and Functional Independence Scale. The patient information form was prepared by the researchers in line with the literature. Permission was obtained from the scale owners for the scales to be used in the study.

Patient Information Form: It was created by the researcher based on the literature. It consists of two parts, individual and disease characteristics of the patients. In the first part; In the second part, individual characteristics such as age, gender, Body Mass Index (BMI), marital status, education level, health insurance, income level, history of surgical intervention, type of surgery and anesthesia applied, toilet habits, gastrointestinal problems, diet, nutrition habits and exercise status, first gas and stool removal time, initiation of oral intake and mobilization status. In the last part of the form, there is a table in which the bowel sounds measured during the patient follow-up will be recorded.

Bristol Stool Scale: The Bristol stool scale will be used to evaluate the individual's first stool.

Forms of feces found on the scale; Type 1 - Goat dung-like, lumpy and chunky hard stool Type 2 - Larger and combined agglomeration Type 3 - Less thick, softer stool with shallow cracks on the surface Type 4 - Stool with a smooth, slippery surface and a soft consistency Type 5 - Pieces of excrement with a consistency to give an edge Type 6 - Soft viscous, more water content, piecemeal stool Type 7 - Hard or soft, watery stool with no solid stool content Gastrointestinal Symptom Rating Scale: It was developed by Revicki et al in 1998 to evaluate common symptoms of gastrointestinal diseases, clinical experience, and views on gastrointestinal symptoms. The scale includes 15 items, each scored on a seven-point Likert-type scale, with values ranging from "no discomfort" to "very severe discomfort". 15 items based on factor analysis; It is divided into five subscales as abdominal pain, reflux, diarrhea, indigestion and constipation. How the individual feels in terms of gastrointestinal problems in the last week is questioned. Higher scores on the scale indicate more severe symptoms. He states that the Cronbach α value in the original scale was between 0.61 and 0.83. In the Turkish adaptation of the scale, the Cronbach Alpha value for all items was found to be 0.82.

General Comfort Scale: It was developed by Kolcaba in 1992 to determine comfort needs and to evaluate the situation of achieving the expected increase in comfort with nursing interventions that provide comfort. The Turkish validity and reliability study of the scale was performed by Kuğuoğlu and Karabacak in 2008. The scale is of a four-point Likert type and contains a total of 48 items. It consists of 3 levels and 4 dimensions. Scale sub-dimensions; relief (16 items), relaxation (17 items) and overcoming problems (15 items). In addition, it is related to physical comfort (12 items), psycho-spiritual comfort (13 items), environmental comfort (13 items) and socio-cultural comfort (10 items). The lowest score that can be obtained from the scale is 48, the median score is 120, and the highest score is 192. As the score obtained from the scale increases, the level of comfort perceived by the patient increases. The original Cronbach Alpha value of the scale was 0.88. In the Turkish adaptation of the scale, the Cronbach Alpha value was found to be 0.83 for all items.

Functional Independence Scale: It is an assessment tool used to evaluate the functional status of individuals. It is divided into two areas: motor and cognitive. It consists of a total of 18 items, 13 in the motor domain and 5 in the cognitive domain. 6 categories and a total of 18 activities are evaluated: self-care (42 points), sphincter control (14 points), transfer (21 points), movement (14 points), communication (14 points) and social perception (21 points). Scale scores range from 18 to 126. A seven point scale is used for each activity. FIM is divided into two measures. Motor FIM consists of 13 functional activities and cognitive FIM consists of 5 cognitive activities. If the total FIM score is 36 points or less, it is defined as high, between 37-72 points as moderate, and 73 points and above as low disability.

Application of Research Patients who meet the sample selection criteria for the study will be informed about the purpose, content and method of the study. This scope of work; Patients who do not defecate in the first 3 days after the surgical intervention will form the experimental and control groups and will be followed by the researcher for 3 days. Experimental and control groups will be determined randomly in patients undergoing surgery who meet the sample selection criteria for the study.

Experimental group

* At the first encounter with the patient; Patient Information Form, Gastrointestinal Symptom Rating Scale, General Comfort Scale and Functional Independence Scale will be applied.
* From the morning of the first day, abdominal massage will be applied to the patients 2 times a day, in the morning and in the evening, for 3 days. Each abdominal massage will be applied for 15 minutes.
* While applying abdominal massage to the patients in the experimental group, the abdominal massage application guidelines (Uysal, Eşer and Akpınar, 2012) in the literature will be used. After each massage application, the patient's bowel sounds/movements will be listened to.
* Medicines such as laxatives, suppositories and enemas will not be given to the experimental group and Bristol Stool Scale will be filled in for patients who defecate within this period.
* In order to evaluate the abdominal massage and its effect on the comfort level of the patients, the Gastrointestinal Symptom Rating Scale, General Comfort Scale and Functional Independence Scale will be applied again at the end of the 3rd day after the application of abdominal massage.

Abdominal Massage Application Guideline:

1. Hands are washed.
2. The healthy/sick individual and their relatives are informed about the procedure.
3. Pain, tenderness, tightness, redness, deterioration of skin integrity and empty bladder are evaluated in the abdominal region of a healthy/sick individual.
4. The healthy/sick individual is placed in the supine position or if there is a risky situation, the bedside of the healthy/sick individual can be 30-45 degrees above.
5. The abdominal region is opened by paying attention to the privacy of the healthy/sick individual. If the skin is damp, it is dried with a towel.
6. A small amount of liquid Vaseline is poured into the hands, and the hands are rubbed to warm the hands and spread the lotion.
7. Superficial effusion is performed by applying light pressure on the abdomen of the healthy/sick individual, starting from the upper epigastric region and downwards, over the iliac bones, from both sides of the pelvis towards the groin. With this effusion, reactive abdominal wall tension due to the first touch is prevented.
8. After the abdominal wall of the healthy/sick individual is relaxed;

   * All movements will be clockwise,
   * Considering the anatomical area starting from the right anterior superior iliac crest, from the level of the ribs to the left anterior superior iliac crest,
   * First of all, massage is applied to the right lower quadrant and right upper quadrant where the ascending colon is located, from the level of the ribs to the left upper quadrant for the transverse colon, and to the left upper and left lower quadrants for the descending colon.
   * The massage applied to each quadrant lasts at least 1 minute and moderate pressure is applied.
9. After the efflorescence movement, the same order is followed and the petrissage movement is performed with the palm.
10. Effeurage and petrissage movements are applied one after the other for 15 minutes, respectively.
11. Finally, vibration is applied using only fingertips for 1 minute and the process is terminated with effusion.
12. The healthy/sick individual is covered and given a comfortable position. Control Group

    * Patients who did not defecate within the first 3 days after surgery will constitute the control group.
    * At the first encounter with the patient; A Patient Information Form, Gastrointestinal Symptom Rating Scale (GSS), General Comfort Scale (GAS) and Functional Independence Scale (FIM) will be administered.
    * From the first encounter, patients will be given medications that are in line with their clinical routine, such as laxatives, suppositories and enemas, according to the doctor's request.
    * Intestinal sounds/movements of the patients will be listened to 6 times, 2 times a day for 3 days.
    * Bristol Stool Scale will be filled in for patients who defecate within this period.
    * At the end of the 3-day follow-up of the patients, Gastrointestinal Symptom Rating Scale, General Comfort Scale and Functional Independence Scale will be applied again and the first stool of the patients who defecate will be evaluated with the Bristol Stool Scale.

Statistical analysis of research data will be done using a package program called SPSS (IBM SPSS Statistics 24).

Institutional permission from Istanbul Medical Faculty and ethics committee approval (Number: E-74555795-050.01.04-412448) from Istanbul University-Cerrahpasa Non-Interventional Research Ethics Committee obtained in order to conduct the study. The expenses of the research will be covered by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and above,
* Being conscious and cooperative,
* Being able to read, write and speak Turkish, not have any cognitive, sensory and spiritual problems,
* Not being pregnant,
* The vital signs are within normal limits after the surgical intervention,
* Failure to defecate for the first 3 days after the surgical intervention,
* Not using pharmacological and non-pharmacological agents with laxative effect after the surgical intervention,
* Continuing inpatient care and treatment in the orthopedics and traumatology clinic for at least 6 days,
* His willingness and volunteering to participate in the study was included.

Exclusion Criteria:

* Be less than 18 years old,
* Not knowing how to read, write and speak Turkish,
* Having any cognitive, sensory and spiritual problems,
* Presence of conditions that prevent the application of abdominal massage (hernia, bowel cancer, history of abdominal surgery and Myocardial Infarction (MI), presence of ileostomy or colostomy and bleeding, etc.),
* Being pregnant
* The vital signs are not within normal limits after the surgical intervention,
* Defecation in the first 3 days after the surgical intervention and using any pharmacological or non-pharmacological agent with laxative effect in this process, Continuing inpatient care and treatment in the orthopedics and traumatology clinic for less than 6 days,
* Not willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Symptom Rating Scale | Change in gastrointestinal symptoms at 6 days
  It is divided into five sub-dimensions: abdominal pain, reflux, diarrhea, indigestion, and constipation. The scale includes 15 items, each scored on a seven-point Likert-type scale, with values ranging from "no discomfort" to "very severe discomfort". Higher scores on the scale indicate more severe symptoms.
General Comfort Scale | Change in comfort level in 6 days
  Evaluates the state of reaching the expected comfort increase result. The scale is scored on a four-point Likert-type scale, each ranging from "strongly agree" to "strongly disagree". The lowest score that can be obtained from the scale is 48, the median score is 120, and the highest score is 192. As the score obtained from the scale increases, the level of comfort perceived by the patient increases.

SECONDARY OUTCOMES:
Functional Independence Scale | Baseline
  It is an assessment tool used to evaluate the functional status of individuals. Self-care (42 points), sphincter control (14 points), transfer (21 points), movement (14 points), communication (14 points) and social perception (21 points) 6 categories and a total of 18 activities are evaluated. Scale scores range from 18 to 126. A 7-point scale is used for each activity. If the total score is 36 points or less, it is defined as high, between 37-72 points as moderate, and 73 points and above as low disability.
Bristol Stool Scale | Up to 6 days after surgery
  It will be used to evaluate the individual's first stool. Forms of feces found on the scale; Type 1 - Goat dung-like, lumpy and chunky hard stool Type 2 - Larger and combined agglomeration Type 3 - Less thick, softer stool with shallow cracks on the surface Type 4 - Stool with a smooth, slippery surface and a soft consistency Type 5 - Pieces of excrement with a consistency to give an edge Type 6 - Soft viscous, more water content, piecemeal stool Type 7 - Hard or soft, watery stool with no solid stool content
Patient Information | Baseline
  It was created by the researcher based on the literature. It consists of two parts, individual and disease characteristics of the patients. In the first part; In the second part, individual characteristics such as age, gender, Body Mass Index (BMI), marital status, education level, health insurance, income level, history of surgical intervention, type of surgery and anesthesia applied, toilet habits, gastrointestinal problems, diet, nutrition habits and exercise status, first gas and stool removal time, initiation of oral intake and mobilization status. In the last part of the form, there is a table in which the bowel sounds measured during the patient follow-up will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Abd-El-Maeboud KHI, Ibrahim MI, Shalaby DAA, Fikry MF. (2009). Gum chewing stimulates early return of bowel motility after caesarean section. BJOG An International Journal of Obstetrics and Gynaecology, 116:1334-1339. 2. Bozkırlı BO, Gündoğdu RH, Ersoy PE, Akbaba S, Temel H, Sayın T. (2012). ERAS protokolü kolorektal cerrahi sonuçlarımızı etkiledi mi? Ulusal Cerrahi Dergisi, 28(3):149-155. doi:10.5152/UCD.2012.05. 3. Çam HH, Nur N.(2015). Hemşirelik ve ebelik öğrencilerinde algılanan stres ile gastrointestinal semptomlar arasındaki ilişki. TAF Preventive Medicine Bulletin, 14(6): 475-482. 4. Çilingir M, Çifter Ç, Kılıçaslan RL. (2004). Mide kanserlerinde ameliyat sonrası erken dönemde enteral ve parenteral beslenme yöntemlerinin morbidite ve mortalite üzerine etkileri. Demet Sağlık Bilimsel Tıp Dergisi, 2(6): 50-54. 5. Herce JL. (2009). Gastrointestinal complications in critically ıll patients: What differs between adults and children? Curr Opin Clin Nutr Metab Care, 12(2): 180-185. 6. Kaçmaz Z, Kaşıkçı M. (2007). Effectiveness of bran supplement in older orthopaedic patients with constipation. Journal of Clinical Nursing, 16(5): 928-936. 7. Kanbir, O. (1998). Klasik Masaj. Bursa: Ekin Kitabevi Yayınları, 189-193. 8. Kaya H, Kaya N, Turan N, Şirin K, Güloğlu S. (2013). Identifying constipation risk in neurosurgery patients. Pielęgniarstwo Neurologiczne iNeurochirurgiczne, 2(3): 96-103. 9. Kolcaba, K. (2003). Comfort Theory And Practice: A vision for holistic health care and research. Springer Publishing Co, New York, 37-58. 10. Kuğuoğlu S, Karabacak, Ü. (2008). Genel Konfor Ölçeğinin Türkçe'ye uyarlanması. Florence Nightingale Hemşirelik Dergisi, 16(61), 16-23. 11. Kyle G. (2008). A proactive approach to the treatment of constipation. Continence, 2(4): 36-44. 12. Kyle, G. (2011). Managing constipation in adult patients. Nurse Prescribing, 9(10): 482-490. 13. Lamas K, Lindholm L, Stenlund H, Engström B, Jacobsson C. (2009). Effects of abdominal massage in management of constipation-A randomized controlled trial. International Journal of Nursing Studies.46(6): 759-767. 14. Lee EY, Mun MS, Lee SH, Cho SM (2011). Perceived stress and gastrointestinal symptoms in nursing students in Korea: A cross sectional survey. BMC Nursing, 10(22): 1-8. 15. McClurg D, Hagen S, Dickinson L. (2011). Abdominal massage for the treatment of constipation. Cochrane Database of Systematic Reviews, 4: 1-5. 16. Perez M, Martinez A. (2009) The Bristol scale - a useful system to assess stool form. Rev Esp EnfermDig. 101(5): 305-311. 17. Resedence TL, Brocklehurst JC. O'Neil PA. (1993). A pilot study on the effect of exercise and abdominal massage on bowel habit in continuing care patients. Clinical Rehabilitation, 7: 204-209. 18. Revicki DA, Wood M, Wiklund I, Crawley J. (1998). Reliability and validity of the gastrointestinal symptom rating scale in patients with gastroesophageal reflux disease. Quality of Life Research, 7: 75-83. 19. Suarez K, Mayer C, Ehlert U, Nater UM. (2010). Psychological stress and self-reported functional gastrointestinal disorders. J Nerv Ment Dis, 198(3): 226-229. 20. Taşdemir N. (2005). Hastaların cerrahi girişim sonrası abdominal distansiyona yönelik deneyimleri. Hacettepe Üniversitesi Sağlık Bilimleri Enstitüsü Cerrahi Hemşireliği, Yüksek Lisans Tezi, Ankara. 21. Tuna N. (2011). A'dan Z'ye Masaj. (6.Baskı). İstanbul: Nobel Tıp Kitabevi, 17-39. 22. Turan N, Asti TA, Kaya N. (2017). Reliability and Validity of the Turkish Version of the Gastrointestinal Symptom Rating Scale. Gastroenterology Nursing, 40(1):47-55. 23. Turan N, Aştı TA, Kaya N. (2017). Nöroşirürji yoğun bakım ünitesinde yatan hastalarda konstipasyon ve hemşirelik bakımı. Hemşirelikte Eğitim ve Araştırma Dergisi, 14 (1): 73-78. 24. Turan N, Aştı TA. (2016). The effect of abdominal massage on constipation and quality of life. Gastroenterology Nursing, 39(1):48-59. 25. Turan N, Aştı T. (2015). Konstipasyon yönetiminde abdominal masajın önemi. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 18(2): 148-154. 26. Ucuzal M, Aldanmaz N. (2015). Genel cerrahi hastalarında ameliyat sonrası konstipasyon riski. İnönü Üniversitesi Sağlık Bilimleri Dergisi, 4 (2): 17-22. 27. Uysal N. (2010). Aralıklı enteral beslenen hastalarda abdominal masajın gastrik rezidüel volüm ve komplikasyonlarına etkisi. Dokuz Eylül Üniversitesi Hemşirelik Yüksekokulu Hemşirelik Esasları Anabilim Dalı, Doktora Tezi, İzmir. 28. Wiesen P, Van Gossum A, Pereiser JC. (2006). Diarrhoea in the critical ill. Current Opinion in Critical Care, 2(2):149-154. 29. Abdominal cerrahi girişim uygulanan hastalarda görülen erken dönem sorunları ve bu sorunlara yönelik hemşirelik uygulamaları. Hacettepe Üniversitesi Sağlık Bilimleri Fakültesi Hemşirelik Dergisi, 2011; 18(2): 36-46. 30. Arı M, Yılmaz E. (2016). Ameliyat öncesi anksiyetenin ameliyat sonrası konstipasyona etkisi. Turk J Colorectal Dis, 2:39-46.
- [Derived] Kucukaydinoglu S, Turan N. The effect of abdominal massage applied after surgery on gastrointestinal symptoms and comfort level. Perioper Med (Lond). 2025 Aug 7;14(1):84. doi: 10.1186/s13741-025-00560-6. PMID 40775370